CLINICAL TRIAL: NCT03810365
Title: Efficacy of Nurse-Delivered Brief Behavioral Treatment to Self-Manage Insomnia in Cancer Survivors
Brief Title: Brief Behavioral Treatment for Insomnia in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Roswell Park Cancer Institute (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Suzanne Dickerson, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002898; 1R01NR018215 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Chronic Insomnia
Keywords: Cancer Survivors; Brief Behavioral Treatment; Older Adults; Attention Control; Intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Brief behavioral treatment for insomnia (Experimental): Brief behavioral treatment for insomnia includes 45 minute individual intervention with two follow up phone calls.
  Interventions: Behavioral: Brief behavioral treatment for insomnia
- Behavioral: Healthy eating control (Active Comparator): Healthy eating control involves a 45 minute individual session with two follow up phone calls.
  Interventions: Behavioral: Healthy Eating Control

INTERVENTIONS:
Behavioral: Brief behavioral treatment for insomnia — Brief Behavioral Treatment for Insomnia includes content on sleep restriction, stimulus control, and sleep hygiene content with 1 month for primary outcome followed by 3 month 12 month follow-up visits.
  Arms: Behavioral: Brief behavioral treatment for insomnia
Behavioral: Healthy Eating Control — Healthy eating control involves healthy eating content with 1 month for primary outcome followed by 3 month and 12 month follow-up visits.
  Arms: Behavioral: Healthy eating control

SUMMARY:
The purpose is to determine whether brief behavioral treatment is effective for insomnia in cancer survivors.

DETAILED DESCRIPTION:
A randomized controlled clinical trial will be used to test the efficacy of this brief behavioral treatment compared to attention control on sleep, mood, functional, status and quality of life and determine predictors for efficacy of Brief Behavioral Treatment for Insomnia (BBTI).

ELIGIBILITY:
Inclusion Criteria:

* > or = 4 weeks from surgery for cancer treatment; chemotherapy and/or radiation therapy; no wait for hormone therapy or targeted treatment for stage I, II, or III: breast, colorectal, prostate, lung cancer
* chronic insomnia

Exclusion Criteria:

* Other preexisting sleep disorders except those with OSA stable on CPAP
* Unstable medical illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne S. Dickerson, PhD, Principal Investigator — University at Buffalo, School of Nursing
Locations (2):
- United States (2):
  - University at Buffalo, Buffalo, New York
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Kwon M, Zhu J, Wilding GE, Larkin K, Gehrman PR, Dickerson SS. Health-related quality of life and mental health outcomes among cancer survivors in an insomnia intervention: a randomized controlled trial. Ann Behav Med. 2025 Jan 4;59(1):kaae096. doi: 10.1093/abm/kaae096. PMID 39887070
- [Derived] Dickerson SS, Kwon M, Wilding GE, Zhu J. Nurse-delivered brief behavioral treatment for insomnia in cancer survivors: a randomized controlled trial. J Cancer Surviv. 2024 Nov 26. doi: 10.1007/s11764-024-01704-1. Online ahead of print. PMID 39589721
- [Derived] Kwon M, Zhu J, Wilding GE, Dickerson SS, Dean GE. Sleep-wake state discrepancy among cancer survivors with insomnia symptoms. Support Care Cancer. 2023 Dec 4;32(1):2. doi: 10.1007/s00520-023-08177-5. PMID 38047967
- [Derived] Kwon M, Dickerson SS, Wilding GE, Aquilina AT, Reid M, Dean GE. A nurse-delivered intervention to reduce insomnia in cancer survivors: Study protocol for a randomized-controlled trial. Contemp Clin Trials. 2022 Nov;122:106939. doi: 10.1016/j.cct.2022.106939. Epub 2022 Sep 28. PMID 36182027
- See also: Dose-response effects of cognitive-behavioral insomnia therapy: a randomized clinical trial. — http://www.ncbi.nlm.nih.gov/pubmed/17326546?dopt=Abstract
- See also: A primary care "friendly" cognitive behavioral insomnia therapy. — http://www.ncbi.nlm.nih.gov/pubmed/12683477?dopt=Abstract
- See also: Effects of a brief behavioral treatment for PTSD-related sleep disturbances: a pilot study. — http://www.ncbi.nlm.nih.gov/pubmed/16777060?dopt=Abstract
- See also: Randomized controlled clinical effectiveness trial of cognitive behavior therapy compared with treatment as usual for persistent insomnia in patients with cancer. — http://www.ncbi.nlm.nih.gov/pubmed/18591549?dopt=Abstract
- See also: How to provide insomnia interventions to people with cancer: insights from patients. — http://www.ncbi.nlm.nih.gov/pubmed/17352006?dopt=Abstract

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a major comprehensive cancer center and ancillary sites in WNY between 6/2019 and 10/2022. The first participant was enrolled 6/6/2019 and last participant was enrolled 9/26/2022. Date of last participant's last visit 11/01/2023.
Pre-assignment Details: Approached for study- n=402, Excluded- n=266 [not meeting inclusion criteria- n=75, Declined to participate- n=47, No response after initial contact- n=144, Total participants completing screening n=136, however, 4 participants quit prior to randomization.
  Final total enrolled participants = 132 with 66 in experimental and 66 in the control group.
Groups:
- Behavioral: Brief Behavioral Treatment for Insomnia: Brief behavioral treatment for insomnia includes 45 minute individual intervention with two follow up phone calls.
  Brief behavioral treatment for insomnia: Brief behavioral Managment of Insomnia content with 1 month 3 month 12 month follow-up visits.
- Behavioral: Healthy Eating Control: Healthy eating control involves a 45 minute individual session with two follow up phone calls.
  Brief behavioral treatment for insomnia: Healthy eating control involves healthy eating content with 1 month 3 month 12 month follow-up visits.
Period: Overall Study
Arm/Group | Behavioral: Brief Behavioral Treatment for Insomnia | Behavioral: Healthy Eating Control
Started | 66 | 66
Completed | 60 | 59
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Behavioral: Brief Behavioral Treatment for Insomnia: Brief behavioral treatment for insomnia includes 45 minute individual intervention with two follow up phone calls.
  Brief behavioral treatment for insomnia: Healthy eating control involves healthy eating content with 1 month 3 month 12 month follow-up visits.
- Total: Total of all reporting groups
Arm/Group | Behavioral: Brief Behavioral Treatment for Insomnia | Behavioral: Healthy Eating Control | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 28 | 70
  >=65 years | 24 | 38 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.26 (11.21) | 65.11 (8.54) | 63.68 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 59 | 58 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 66 | 132
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — the Insomnia Severity Index is a self report brief screening tool with seven items that asks respondents to rate the nature and symptoms of their sleep problems and the degree to which insomnia interferes with daily functioning and overall distress created by sleep problems using a likert type scale. Scores from 8-14 meaures subthreshhold insomnia, 15-21 measures moderate insomnia, and 22-28 measures severe insomnia. Higher scores reflect worse outcomes.
  units on a scale | 12.56 (3.61) | 14.26 (4.33) | 13.41 (4.06)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index
Description: One month after the intervention, experimental group mean for Insomnia Severity Index will be compared to control group mean Insomnia Severity Index.
  The Insomnia Severity Index is a self report brief screening tool with seven items that asks respondents to rate the nature and symptoms of their sleep problems and the degree to which insomnia interferes with daily functioning and overall distress created by sleep problems using a likert type scale Scores between 0-7 have no clinically significant insomnia. Scores between 8-14 have sub threshold insomnia. Scores between 15-21 have moderate clinical insomnia. Scores between 22-28 have severe clinical insomnia.
Time Frame: one month
Population: The main efficacy was determined at one month after the intervention. The study continued with measurements at 3 months and 12 months to determine durability. additional participants dropped out and the final numbers in the study were 60 experimental and 59 control.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Behavioral: Brief Behavioral Treatment for Insomnia: Brief behavioral treatment for insomnia intervention includes 45 minute individual intervention with two follow up phone calls.with 1 month followup for Insomnia Severity Index measure
- Behavioral: Healthy Eating Control: Healthy eating control involves a 45 minute individual session with two follow up phone calls with one month followup for Insomnia severity Index measure.
Arm/Group | Behavioral: Brief Behavioral Treatment for Insomnia | Behavioral: Healthy Eating Control
Number analyzed (Participants) | 62 | 60
score on a scale | 7.03 [5.78 to 8.28] | 9.26 [7.90 to 10.62]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Behavioral: Brief Behavioral Treatment for Insomnia | Behavioral: Healthy Eating Control
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/60
Other Adverse Events (participants affected / at risk) | 0/62 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT03810365/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT03810365/ICF_001.pdf